CLINICAL TRIAL: NCT04074044
Title: Evaluation of a New Bladder Health Mobile Application in Pregnancy
Acronym: BHmApp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Elie Mulhem, Vice Chair, Department of Family Medicine and Community Health, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-157
Record Dates: First submitted 2019-08-27; First posted 2019-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence
Keywords: Prevention; Pregnancy; Mobile Health App; PEMAT questionnaire
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Single group, open label evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BHmApp users (Experimental): Participants using BHmApp tor bladder education and training
  Interventions: Behavioral: BHmApp

INTERVENTIONS:
Behavioral: BHmApp — Use of BHmApp for bladder education and training in pregnancy

SUMMARY:
Millions of women experience involuntary loss of urine called urinary incontinence (UI). UI can be slightly bothersome or totally debilitating. Women experience UI twice as often as men. Urinary incontinence can also be a persistent condition caused by underlying physical problems or changes, including pregnancy and childbirth. UI symptom severity progress dynamically and are also sustained over time. High quality evidence shows that pelvic floor muscle training (PFMT) during pregnancy effectively reduces the risk of UI during pregnancy and the postpartum period. There is a critical need for a low cost and easily accessible program to prevent UI in pregnancy and postpartum that can reach a large number of women. A mobile health application that teaches UI preventive program during pregnancy has the potential of being a cost effective tool to reach a large number of pregnant women. The Bladder Health Mobile Application (BHmApp) will teach pregnant women new habits and exercises that will keep their bladder healthy during pregnancy and decrease the risk of UI during this period of a woman's life that is considered high risk for developing UI. In this pilot study, it is proposed to evaluate the understand and effectively use the BHmApp, and the feasibility of using the BHmApp during pregnancy.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is the involuntary and unintentional leaking of urine. Over 20 million of women experience UI, approximately 34% (range 25-45%) of all US women are affected indicating a significant healthcare concern with both financial and quality of life implications. The financial cost of UI in the United States (U.S) exceeds $65 billion per year (in year 2007 dollars), and it is projected that the cost will be $82.6 billion in 2020.Women with UI feel shame about this condition, report poor self-esteem, and are at increased risk of depression. Pregnancy is a high-risk time for developing stress UI, urine leakage with physical effort, with a reported prevalence of 35-67% during pregnancy and 31% postpartum. Pregnancy also places women at increased risk of developing UI later in life.

High quality evidence shows that pelvic floor muscle training (PFMT) during pregnancy effectively reduces the risk of UI during pregnancy and the postpartum period by 39-59%. A recent Cochrane review examined the evidence for PFMT based on 38 trials involving 9,892 women from 20 countries. The authors concluded that in continent pregnant women, performing antenatal PFMT may decrease the risk of UI in late pregnancy and in the mid-postnatal period greater 3 to six months postpartum. However, evidence shows that many women in the U.S. do not receive effective PFMT. PFMT to prevent UI is not routinely offered or well taught to pregnant women.

There is a critical need for a low cost and easily accessible program to prevent UI in pregnancy and postpartum that can reach a large number of women. Such a program could reduce the financial and psychological impact of UI on pregnant women, lower the risk of UI with its associated negative outcomes and address a priority area identified by National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK). A mobile health application that teaches UI preventive program during pregnancy has the potential of being a cost effective tool to reach a large number of pregnant women. The plan is to offer PFMT, the Knack (squeeze before you sneeze trick), bladder training (BT) with urge suppression and healthy bladder education (fluid modification, bowel habits) using a mobile health application that allows women to learn and practice these new habits anytime and anywhere that is convenient to them. In the pilot studies, as supported by other studies, it was learned that the main obstacles to preventing UI by means of PFMT are the feasibility of group classes and low adherence to the exercise routine. Mobile health application (mApp) offers an innovative approach to improve feasibility. PFMT mApps showed effectiveness in women with stress UI and improved adherence to PFMT in women with UI. Additionally, stress UI self-management that includes PFMT with mApp has been shown to be cost-effective. Measurement of adherence to behavioral protocols has often been overlooked in research. Few studies provide information about how adherent women were with PFMT and the literature is sparse on methods to identify barriers and improve adherence. Adherence to PFM exercises during pregnancy was reported to be between 16%-69%, and adherence rates 4-6 weeks after delivery were 43%-83%. Common reasons for not doing PFMT during pregnancy and postpartum include exercises are: forgetting, being too busy, and the belief they have become unnecessary due to the absence of symptoms. Using a mobile App is an innovative way to address these obstacles. To help women overcome these particular barriers, this study proposes a Bladder Health mobile application (BHmApp) that will use various forms of reminders, provide exercise aids, link daily exercises to environmental cues, and integrate exercises into the patient's everyday activities.

To support adherence, the BHmAPP will communicate realistic expectations, make it clear that it may take weeks to months for symptom improvement, and it may be irregular, with "good" days and "bad" days. The BHmApp can provide support by tracking and reinforcing progress, identifying and addressing barriers, and encouraging persistence.

During the last year, the team worked on designing and building the BHmApp aimed to teach pregnant women new habits and exercises that will keep their bladder healthy during pregnancy and decrease the risk of UI during this period of a woman's life that is considered high risk for developing UI. In this pilot study, it is proposed to evaluate the ability to comprehend the tool and take appropriate actions using the BHmApp, and the feasibility of using the BHmApp during pregnancy.

The BHmApp is designed to: effectively engage pregnant women prior to development of UI and associated bladder symptoms, teach them new health habits that will decrease their risk of UI and associated bladder symptoms and increase their ability to keep their bladder healthy. The proposed project is innovative in the following ways:

1. BHmApp focus is the prevention of UI. Currently, there are many mApps that teach PFMT to treat UI, most use simple instruction protocols, use the same protocol for all patients, and end up working the same way as simple verbal instruction. This BHmApp protocol is designed for pregnant women, offering training for PFMT, Knack, BT and urge suppression and bladder health strategies, allows women to connect with a bladder health coach to ask questions, offers notification reminders of exercise time, and a way for women to record and track adherence to PFMT.
2. The BHmApp is built specifically for pregnant women. With pregnancy being the high-risk time in a woman's life to develop UI, there is a need for a UI prevention program that can reach large numbers of women at low cost. The BHmApp is designed to teach pregnant women these new habits and skills, and offers a new opportunity in the effort to prevent UI. This BHmApp takes into consideration the physiologic changes in a woman's body during pregnancy, and the restrictions to certain exercises and habits during pregnancy. For example, bladder health is not practiced until 4 weeks after delivery and PFMT is done in sitting position after 20-weeks gestation.
3. The BHmApp format allows participants to access the health information at any time, and anywhere that is convenient for them. Pregnancy is a busy period of time in a woman's life, with increased healthcare visits, preparing for new baby, and an increased chance of fatigue and insomnia. Offering a chance to gain new knowledge and learn new habits through short (2-3 minutes) lessons, that can be accessed at a woman's convenience, would significantly increase the chances of learning these important skills and habits during pregnancy.

   Participants will complete the following study activities:

   Study Initiation:

   • Complete demographics questionnaire (name, medical Record Number (MRN), email address, Tel. No. Cell Phone Carrier)
   * Complete International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) - measures UI frequency, severity, and impact on Quality of Life (QOL)
   * Download the Bladder Health Mobile Application (BHmApp) on phone

     4 Weeks after BHmApp Download or at End of App Lessons:
   * Complete the Patient Education Materials Assessment Tool (PEMAT) - (about 22-24 weeks gestation) - a scoring questionnaire to assess understandability and actionability for audiovisual or printed patient education materials.

   26-28 Weeks Gestation Email/Text Sent • Complete Pelvic Floor Muscle Training (PFMT) adherence questionnaire

   30-32 Weeks Gestation Email/Text Sent • Complete Pelvic Floor Muscle Training (PFMT) adherence questionnaire

   34-36 Weeks Gestation Email/Text Sent

   • Complete Pelvic Floor Muscle Training (PFMT) adherence questionnaire
   * Complete International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF)

     6 Weeks Postpartum Email/Text Sent
   * Complete International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF)
   * Complete Pelvic Floor Muscle Training (PFMT) adherence questionnaire and Bladder Training (BT) adherence questionnaire

     12 weeks Postpartum Email/Text Sent
   * Complete International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF)
   * Complete Pelvic Floor Muscle Training (PFMT) adherence questionnaire and Bladder Training (BT) adherence questionnaire

   The BHmApp is 2-4 minutes in length with separate quick and slow exercises. Soft music is played through the entire recording with the sound slightly increasing during the relaxation period. The work-out music is motivational but not too fast.

   The app contains 3 audio lessons:

   Lesson 1, the quick squeeze Lesson 2, the slow squeeze Lesson 3, practice a full set of a pelvic muscle exercises including the quick squeeze and slow squeeze

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women age 18 years or older at 10-18 weeks gestation
* Ability to understand English
* Negative history or no more than 5 episodes of UI in the past 12 months
* Negative history of neuromuscular or genitourinary conditions
* Low-risk antepartum
* Singleton pregnancy
* Owner of a smart phone

Exclusion Criteria:

• High-risk pregnancy, including medical complications during pregnancy, such as preterm delivery, preterm premature rupture of membranes, diabetes, or hypertensive disorders and history of prior diagnosis or treatment (behavioral, drug or surgical) for urinary incontinence

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Understandability score from Patient Education Materials Assessment Tool (PMAT) questionnaire | 4 weeks after enrollment
  Percentage of positive responses to understandability questions (1-19) of the PMAT survey, where each question has a score of 0=disagree and 1=agree for each question. The sum of total points is divided by the sum of total possible points and multiplied by 100 to get percentage. A high score indicates the participant understood the material well.
Actionability score from Patient Education Materials Assessment Tool (PMAT) questionnaire | 4 weeks after enrollment
  Percentage of positive responses to actionability questions (20-26) of the PMAT survey, where each question has a score of 0=disagree and 1=agree for each question. The sum of total points is divided by the sum of total possible points and multiplied by 100 to get percentage. A high score indicates the participant was able to develop an action plan from the material.

SECONDARY OUTCOMES:
Recruitment Success | At enrollment
  Percentage of patients enrolled of all those approached for study
Retention rate | 12 weeks postpartum
  Number of participants who remain enrolled in the study through 12 weeks postpartum.
Data completion rate | 12 weeks post partum
  Number of participants who return completed study questionnaire 12 weeks post partum
Urinary Incontinence (UI) rate - baseline | at enrollment
  Number of participants scoring mild, moderate, severe or very severe incontinence on the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), a 3-question scale measuring UI frequency, severity and impact on quality of life with a maximum possible score of 21. 1-5 is considered mild incontinence, a score of 6-12 is considered moderate incontinence, 13-18 is considered severe incontinence and 19-21 very severe incontinence.
Urinary Incontinence (UI) rate - 34-36 weeks gestation | 34-36 weeks gestation
  Number of participants scoring mild, moderate, severe or very severe incontinence on the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), a 3-question scale measuring UI frequency, severity and impact on quality of life with a maximum possible score of 21. 1-5 is considered mild incontinence, a score of 6-12 is considered moderate incontinence, 13-18 is considered severe incontinence and 19-21 very severe incontinence.
Urinary Incontinence (UI) rate - 6 weeks postpartum | 6 weeks post partum
  Number of participants scoring mild, moderate, severe or very severe incontinence on the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), a 3-question scale measuring UI frequency, severity and impact on quality of life with a maximum possible score of 21. 1-5 is considered mild incontinence, a score of 6-12 is considered moderate incontinence, 13-18 is considered severe incontinence and 19-21 very severe incontinence.
Urinary Incontinence (UI) rate - 12 weeks postpartum | 12 weeks post partum
  Number of participants scoring mild, moderate, severe or very severe incontinence on the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF), a 3-question scale measuring UI frequency, severity and impact on quality of life with a maximum possible score of 21. 1-5 is considered mild incontinence, a score of 6-12 is considered moderate incontinence, 13-18 is considered severe incontinence and 19-21 very severe incontinence.
Adherence to Pelvic Floor Muscle Training (PFMT) - 26-28 weeks gestation | 26-28 weeks gestation
  Sum of score on questions 1-4 of the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire. The maximum score is 21 with a higher score indication greater adherence to pelvic floor exercises.
Adherence to Pelvic Floor Muscle Training (PFMT) - 30-32 weeks gestation | 30-32 weeks gestation
  Sum of score on questions 1-4 of the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire. The maximum score is 21 with a higher score indication greater adherence to pelvic floor exercises.
Adherence to Pelvic Floor Muscle Training (PFMT) - 34-36 weeks gestation | 34-36 weeks gestation
  Sum of score on questions 1-4 of the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire. The maximum score is 21 with a higher score indication greater adherence to pelvic floor exercises.
Adherence to Pelvic Floor Muscle Training (PFMT) - 6 weeks postpartum | 6 weeks postpartum
  Sum of score on questions 1-4 of the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire. The maximum score is 21 with a higher score indication greater adherence to pelvic floor exercises.
Adherence to Pelvic Floor Muscle Training (PFMT) - 12 weeks postpartum | 12 weeks postpartum
  Sum of score on questions 1-4 of the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire. The maximum score is 21 with a higher score indication greater adherence to pelvic floor exercises.
Bladder Training Adherence - 6 weeks postpartum | 6 weeks post partum
  Number of patients indicating "yes" to the bladder training adherence question of the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire. A positive response indicates bladder training was used.
Bladder Training Adherence - 12 weeks postpartum | 12 weeks post partum
  Number of patients indicating "yes" to the bladder training adherence question of the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire. A positive response indicates bladder training was used.
Voiding interval - 6 weeks postpartum | 6 weeks post partum
  Change in estimated number of minutes between urinations after completing bladder training, as reported on the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire.
Voiding interval - 12 weeks postpartum | 12 weeks post partum
  Change in estimated number of minutes between urinations after completing bladder training, as reported on the Pelvic Floor Muscle Exercise and Bladder Training Adherence questionnaire.
Barriers to Use of bladder training - 6 weeks postpartum | 6 weeks post partum
  Numbers of patients reporting each of 4 possible reasons as barriers to use of bladder training: Average time between urinations was as recommended, it was too complicated to fit into daily life, it was not a technique the participant wanted to try, or other.
Barriers to Use of bladder training - 12 weeks postpartum | 12 weeks post partum
  Numbers of patients reporting each of 4 possible reasons as barriers to use of bladder training: Average time between urinations was as recommended, it was too complicated to fit into daily life, it was not a technique the participant wanted to try, or other.

CONTACTS AND LOCATIONS:
Overall Officials: Elie Mulhem, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospitals, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No pan to share individual patient data